CLINICAL TRIAL: NCT03120247
Title: Pharmacokinetics and Pharmacodynamics of Three Doses of Oral Trans-mucosal Dexmedetomidine for Premedication in Patients Undergoing Modified Radical Mastectomy
Brief Title: Pharmacokinetics and Pharmacodynamics of Oral Transmucosal Dexmedetomidine.
Acronym: OTM/DEX/PK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Assistant professor in anesthesia and intensive care, Faculty of medicine, Assiut university, Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IORG0006563/no. 377
Record Dates: First submitted 2017-04-05; First posted 2017-04-19 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic and pharmacodynamic study of three different doses of oral transmucosal dexmedetomidine
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- DEX I (Active Comparator): OTM Dexmetetomidine 1µg/kg Oral transmucosal dexmedetomidine pharmacologically prepared as a jel substance will be administered to the buccal mucosa 30 mins before the operative procedure.
  Interventions: Drug: OTM Dexmedetomidine 1µg/ kg.
- DEX II (Active Comparator): OTM Dexmetetomidine0.75µg/kg Oral transmucosal dexmedetomidine pharmacologically prepared as a jel substance will be administered to the buccal mucosa 30 mins before the operative procedure.
  Interventions: Drug: OTM Dexmedetomidine 0.75µg/ kg.
- DEX III (Active Comparator): OTM Dexmetetomidine 0.5µg/kg. Oral transmucosal dexmedetomidine pharmacologically prepared as a jel substance will be administered to the buccal mucosa 30 mins before the operative procedure.
  Interventions: Drug: OTM Dexmedetomidine 0.5µg/ kg.

INTERVENTIONS:
Drug: OTM Dexmedetomidine 1µg/ kg. — Oral transmucosal dexmedetomidine pharmacologically prepared as a jel substance will be administered to the buccal mucosa 30 mins before the operative procedure.
  Other Names: Precedex
  Arms: DEX I
Drug: OTM Dexmedetomidine 0.75µg/ kg. — Oral transmucosal dexmedetomidine pharmacologically prepared as a jel substance will be administered to the buccal mucosa 30 mins before the operative procedure.
  Other Names: Precedx
  Arms: DEX II
Drug: OTM Dexmedetomidine 0.5µg/ kg. — Oral transmucosal dexmedetomidine pharmacologically prepared as a jel substance will be administered to the buccal mucosa 30 mins before the operative procedure.
  Other Names: Precedex
  Arms: DEX III

SUMMARY:
Oral trans-mucosal administration is relatively easy and convenient, it also reduces first pass metabolism and has been used successfully for fentanyl, ketamine, and midazolam premedication.

DETAILED DESCRIPTION:
The alpha2-adrenoceptor agonist, dexmedetomidine, was originally developed as a sedative and analgesic drug for use in intensive care. However, it has a number of unique pharmacodynamic properties, which also make it useful in anesthesia including; decreased MAC, analgesia without respiratory depression and a significant reduction in catecholamine secretion. Also it has been used off-label as an adjunctive agent for sedation and analgesia in patients in the critical care unit and for sedation during non-invasive procedures in radiology. It also has a potential role as part of anesthesia care to prevent emergence delirium and post-anesthesia shivering.

Oral trans-mucosal administration is relatively easy and convenient, it also reduces first pass metabolism and has been used successfully for fentanyl, ketamine, and midazolam premedication.

The current literature is focused in studying the sedative and analgesic effects of intravenously administered dexmedetomidine. Pharmacodynamics and pharmacokinetic studies undertaken on alternative routes of dexmedetomidine administration are lacking. The pharmacokinetic properties of trans-mucosal administration of dexmedetomidine have been demonstrated in one study only, and the clinical effects of non-parenteral administration of dexmedetomidine have been described in anecdotal case reports.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I - II.
* Aged between 20 and 60 years.
* Scheduled for modified radical mastectomy

Exclusion Criteria:

* Cardiac disease.
* Hepatic disease.
* Renal disease.
* History of alcohol or drug abuse.
* Patients with a known allergy to the study drug

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 360 minutes.
  Two milliliters of blood will be collected for determination of Peak Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Sedation preoperative | 30 minutes
  Sedation score is recorded pre-operatively every 5minutes for 30 minutes after OTM DEX administration
Blood pressure preoperative | 30 minutes.
  Non invasive blood pressure will be recorded every 5 minutes for 30 minutes after OTM DEX administration.
Heart rate preoperative | 30 minutes
  Heart rate will be recorded every 5 minutes for 30 minutes after OTM DEX administration.
Area under the plasma concentration versus time curve (AUC) | 360 minutes.
  Two milliliters of blood will be collected for determination of Area under the plasma concentration versus time

CONTACTS AND LOCATIONS:
Overall Officials: Saher A Mohamed, MD, Principal Investigator — Assistant professor in anesthesia and pain management, South Egypt Cancer Institute, faculty of medicine, Assiut university.
Locations (1):
- South Egypt cancer institute, Assiut university, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamed SA, Abdel-Ghaffar HS, Hassan NA, El Sherif FA, Shouman SA, Omran MM, Hassan SB, Allam AAAE, Sayed DG. Pharmacokinetics and Pharmacodynamics of 3 Doses of Oral-Mucosal Dexmedetomidine Gel for Sedative Premedication in Women Undergoing Modified Radical Mastectomy for Breast Cancer. Anesth Analg. 2021 Feb 1;132(2):456-464. doi: 10.1213/ANE.0000000000005108. PMID 32889844